CLINICAL TRIAL: NCT00767195
Title: Power Spectral Analysis of Lung Sounds Detected at Bilateral Lung Bases in Patients With Cardiogenic and Non-cardiogenic Pulmonary Edema
Brief Title: Power Spectral Analysis of Breath Sound in Pulmonary Edema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Cheng-Deng Kuo, MD, PhD, Professor, Taipei Veterans General Hospital
Other Study IDs: VGHIRB97-01-02A; 200808065R
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Pulmonary Edema
Keywords: pulmonary edema; cardiogenic; non-cardiogenic; mortality; length of stay
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1. Control group: Patients in the intensive care unit who have no pulmonary edema
- 2. Study group 1: Patients with cardiogenic pulmonary edema in the intensive care unit
- 3. Study group 2: Patients with non-cardiogenic pulmonary edema in the intensive care unit

SUMMARY:
Pulmonary edema can be classified into "cardiogenic pulmonary edema" and "non-cardiogenic pulmonary edema" according to the underlying etiology. Cardiogenic pulmonary edema is caused by the dysfunction in the cardiac pumping capability, leading to the transudation accumulation in the pulmonary peri-capillary space. The predisposing factors of non-cardiogenic pulmonary edema are numerous, including severe infection, renal failure, auto-immun reaction, etc. The mortality rate of pulmonary edema is relatively high, especially the non-cardiogenic one. To distinguish the type of pulmonary edema at the early stage is important for its treatment.

Lung sound analysis via stethoscope is a simple diagnostic method to lung diseases clinically. Among many kinds of lung sounds, the "crackle" and "rale" are frequently found in pulmonary edema. "Rale" is also called "moist rale". It is considered as low-frequency wheezes and is often seen in cardiogenic pulmonary edema. On the other hand, "crackle" is also called "dry rale", which is a kind of high-frequency wheezes and usually seen in Acute Respiratory Distress Syndrome (ARDS) that is classified into non-cardiogenic pulmonary edema.

This proposed project intends to establish a digital diagnostic method for pulmonary edema. The lung sound of patient with pulmonary edema will be collected by the lung sound acquisition system. By identifying the significant spectrum characteristics of cardiogenic pulmonary edema and non-cardiogenic pulmonary edema, the diagnostic system might be established.

DETAILED DESCRIPTION:
Pulmonary edema is caused by the disorder of liquid accumulation between lung capillary and peri-capillary tissue. This lung disease can be classified into "Cardiogenic pulmonary edema" and "Non-cardiogenic pulmonary edema" according to the underlying etiology. Cardiogenic pulmonary edema is caused by the dysfunction in the cardiac pumping capability, leading to the transudation accumulation in the pulmonary peri-capillary space. Pulmonary ventilation and perfusion mismatch developed and shortness of breath ensued. The predisposing factors of non-cardiogenic pulmonary edema are numerous, including severe infection, renal failure, auto-immun reaction, etc. The mortality rate of pulmonary edema is relatively high, especially the non-cardiogenic one. To distinguish the type of pulmonary edema at the early stage is important for its treatment.

Stethoscopes are widely used in clinical diagnosis in different diseases. Lung sound analysis via stethoscope is a simple diagnostic method to lung diseases clinically. Among many kinds of lung sounds, the "crackle" and "rale" are frequently found in pulmonary edema. "Rale" is also called "moist rale". It is considered as low-frequency wheezes and is often seen in cardiogenic pulmonary edema. On the other hand, "crackle" is also called "dry rale", which is a kind of high-frequency wheezes and usually seen in Acute Respiratory Distress Syndrome (ARDS) that is classified into non-cardiogenic pulmonary edema.

By simply listening to the lung sounds, a doctor can determine whether the patient has pulmonary edema or not, and whether the pulmonary edema if present is cardiogenic or not. This listening diagnostic method is simple and non-invasive. However, its accuracy is limited by such factors as the doctor's subjectiveness and interference from other physiological signals. Also, it is sometimes difficult to distinguish cardiogenic pulmonary edema from non-cardiogenic pulmonary edema just by auscultation only. Advanced diagnostic method (such as echocardiography) is often needed for further evaluation of lung problems.

This proposed project intends to establish a digital diagnostic method for pulmonary edema by integrating the medical expertise and resources of NTUH (National Taiwan University Hospital) and the engineering ability of NCU-EE (Department of Electrical Engineering, National Central University) in computer, electronics, and signal processing. We will apply the developed tool to lung sound acquisition hardware system for pulmonary edema diagnosis and set up an electronic diagnostic system. The lung sound of patient with pulmonary edema will be collected by this lung sound acquisition hardware system for the establishment of a Pulmonary Edema Library. By identifying the significant spectrum characteristics of cardiogenic pulmonary edema and non-cardiogenic pulmonary edema, the diagnostic system might be established.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the intensive care unit using ventilator

Exclusion Criteria:

* Asthma, COPD, non-ventilated patients

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without pulmonary edema (control group), with cardiogrnic edema (study group 1) and non-cardiogrnic edema (study group 2)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Low-Tone Ho, MD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Intensive Care Unit, Taipei, Taiwan